CLINICAL TRIAL: NCT02579915
Title: Phase 2 Randomized Controlled Trial of Attention and Interpretation Modification (AIM) for Anxiety Disorders in Primary Care
Brief Title: Developing a Low-Intensity Primary Care Intervention for Anxiety Disorders (AIM-PC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Mclean Hospital (Other); Memorial Hospital of Rhode Island (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Courtney Beard, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1308000908-Phase 2; 1R34MH097820-01A1 (NIH)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FaceAnxiety - Mental Habits (Experimental): Treatment will consist of 8, 30-minute, twice-weekly sessions designed to: a) decrease attention bias to threat and b) extinguish threat interpretations/reinforce benign interpretations of ambiguity. Attention bias will be modified via a dot probe task that increases attentional control by directing attention away from threat faces via probe location. Patients will complete 256 trials per session. Interpretation bias will be modified via a word-sentence association task which provides positive feedback when participants endorse benign interpretations of ambiguous sentences and negative feedback for threat interpretations. Participants will complete 150 training trials per session. A FaceAnxiety Specialist facilitates program completion.
  Interventions: Behavioral: FaceAnxiety; Behavioral: Symptom Tracking
- FaceAnxiety - Symptom Tracking (Active Comparator): Treatment will consist of weekly self-assessment of anxiety and depression symptoms via on-line surveys. A FaceAnxiety Specialist will facilitate program completion.
  Interventions: Behavioral: Symptom Tracking

INTERVENTIONS:
Behavioral: FaceAnxiety — Computerized treatment targeting mental habits and primary care linkage.
  Other Names: Cognitive Bias Modification
  Arms: FaceAnxiety - Mental Habits
Behavioral: Symptom Tracking — Weekly self-assessment with validated questionnaires and primary care linkage

SUMMARY:
The purpose of the study is to develop a personalized, user-friendly computerized treatment for anxiety disorders linked to primary care. The computerized treatment is a type of Cognitive Bias Modification, which targets attention and interpretation biases known to maintain anxiety disorders.

DETAILED DESCRIPTION:
The primary goals of our 3-year, 2-phase project are to develop AIM for primary care linkage and assess its feasibility and acceptability. This protocol description only pertains to Phase 2 (Randomized Controlled Trial).

42 primary care patients with primary Generalized Anxiety Disorder, Social Anxiety Disorder, and/or Panic Disorder (with or without Agoraphobia) will be randomly assigned to the AIM treatment or to a symptom tracking control group. Full assessments will occur pre- and post-treatment and 3-months follow-up. A mid-treatment assessment will include measures of cognitive biases and the primary outcome. Weekly measures of anxiety and depression will be collected, as will feedback from patients and PCPs about the research and delivery procedures.

ELIGIBILITY:
Inclusion Criteria:

Study site patient Age ≥18 Primary diagnosis of Generalized anxiety disorder (GAD), Social Phobia (SP), and/or panic disorder with or without agoraphobia (PD/A) At least moderate anxiety severity (GAD-7 score > 10) English-speaking If on psychopharmacotherapy, stable dose for 3 months; to minimize learning effects, patients taking benzodiazepines will complete AIM prior to their first dose of the day No current psychotherapy No current severe psychiatric symptoms requiring immediate attention (e.g., imminent suicidality, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa B Weisberg, PhD, Principal Investigator — Brown University; Courtney Beard, PhD, Principal Investigator — Harvard Medical School/McLean Hospital
Locations (1):
- Family Care Center at Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FaceAnxiety - Mental Habits | FaceAnxiety - Symptom Tracking
Started | 19 | 21
Completed | 9 | 16
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Population: Note that one participant in each arm did not provide age data. Thus, total number of baseline participants differs from those analyzed for age.
Groups:
- Total: Total of all reporting groups
Arm/Group | FaceAnxiety - Mental Habits | FaceAnxiety - Symptom Tracking | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant from each arm did not provide their age. These data are missing.
  Participants
    number analyzed (Participants) | 18 | 20 | 38
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 18 | 35
    >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Note that one participant in each arm did not provide age data. Thus, total number of baseline participants differs from those analyzed for age.
  years
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 42.6 (14.16) | 41.1 (15.88) | 42.1 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in the symptom monitoring arm did not provide their sex on the demographic form. This data is missing.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Female | 14 | 16 | 30
    Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 14 | 8 | 22
  Unknown or Not Reported | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 14 | 13 | 27
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Rating Scale
Description: Number of participants who achieved a 20% reduction in their interview-administered Hamilton Anxiety Rating Scale Total Score.
Time Frame: 6-8 weeks after first treatment session
Population: We only analyzed participants who completed their post-treatment assessment, which is required to calculate their % reduction in symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | FaceAnxiety - Mental Habits | FaceAnxiety - Symptom Tracking
Number analyzed (Participants) | 8 | 16
Participants | 5 | 6

2. Secondary Outcome: 7-item Generalized Anxiety Disorder Scale
Time Frame: 6-8 weeks after first treatment session
Reporting Status: Not Posted

3. Secondary Outcome: Patient Health Questionnaire-9
Time Frame: 6-8 weeks after first treatment session
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were followed for 3 months following their post-treatment assessment. Thus, in total participants were followed for up to 6 months depending on how quickly they completed the treatment.
Arm/Group | FaceAnxiety - Mental Habits | FaceAnxiety - Symptom Tracking
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FaceAnxiety - Mental Habits (N=19) | FaceAnxiety - Symptom Tracking (N=21)
suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02579915/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02579915/SAP_001.pdf